CLINICAL TRIAL: NCT02112903
Title: Interventional, Randomised, Double-blind 4-way Crossover Study Comparing the Gastro-intestinal Tolerability and Absorption Profile of Vortioxetine After Administration of Modified-release Formulations and Immediate-release Formulation in Healthy Women
Brief Title: Study Comparing the Gastro-intestinal Tolerability and Absorption Profile of Vortioxetine After Administration of Modified-release Formulations and Immediate-release Formulation in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15947A; 2014-000121-20 (EudraCT Number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Encapsulated vortioxetine IR tablet, 20 mg (Experimental): Single oral dose
  Interventions: Drug: Encapsulated vortioxetine IR tablet, 20 mg
- Vortioxetine MR capsule 20 mg (pH 5.5) (Experimental): Single oral dose
  Interventions: Drug: Vortioxetine MR capsule 20 mg (pH 5.5)
- Vortioxetine MR capsule 20 mg (pH 6.0) (Experimental): Single oral dose
  Interventions: Drug: Vortioxetine MR capsule 20 mg (pH 6.0)
- Vortioxetine MR capsule 20 mg (pH 7.0) (Experimental): Single oral dose
  Interventions: Drug: Vortioxetine MR capsule 20 mg (pH 7.0)

INTERVENTIONS:
Drug: Encapsulated vortioxetine IR tablet, 20 mg
  Arms: Encapsulated vortioxetine IR tablet, 20 mg
Drug: Vortioxetine MR capsule 20 mg (pH 5.5)
  Arms: Vortioxetine MR capsule 20 mg (pH 5.5)
Drug: Vortioxetine MR capsule 20 mg (pH 6.0)
  Arms: Vortioxetine MR capsule 20 mg (pH 6.0)
Drug: Vortioxetine MR capsule 20 mg (pH 7.0)
  Arms: Vortioxetine MR capsule 20 mg (pH 7.0)

SUMMARY:
The purpose of this study is to evaluate the gastro-intestinal tolerability (nausea, vomiting, diarrhoea, abdominal discomfort, and abdominal pain) of vortioxetine following single oral doses of three modified-release (MR) capsules with differently coated multiple particles compared to one immediate-release (IR) tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ≥18 and ≤45 years of age with a body mass index (BMI) of >18.5 and <30.0 kg/m2.
* Women will be of child-bearing potential with a confirmed non-pregnant and non-lactating status.

Other protocol-defined Inclusion and Exclusion Criteria may apply.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal tolerability (nausea) measured with 11-point Numerical Rating Scale | Up to 24 hours post-dose in each treatment period
Gastro-intestinal tolerability (abdominal pain) measured with 11-point Numerical Rating Scale | Up to 24 hours post-dose in each treatment period
Gastro-intestinal tolerability (abdominal discomfort) measured with 11-point Numerical Rating Scale | Up to 24 hours post-dose in each treatment period
Frequency, severity and duration of reported gastro-intestinal tolerability (nausea, vomiting, diarrhoea, abdominal discomfort and abdominal pain) | Up to 72 hours post-dose in each treatment period
Area under the vortioxetine plasma concentration-time curve from zero to 72 hours post-dose (AUC0-72h) | Up to 72 hours postdose
Maximum observed concentration (Cmax) of vortioxetine | Up to 72 hours postdose
Nominal time corresponding to the occurrence of Cmax (tmax) | Up to 72 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- GB801, London, United Kingdom